CLINICAL TRIAL: NCT04047654
Title: Efficacy and Safety of Oral Anticoagulants Among Thai Octogenarians With Nonvalvular Atrial Fibrillation : A Retrospective Study
Brief Title: Efficacy and Safety of Oral Anticoagulants Among Thai Octogenarians With Nonvalvular Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: NOACs in Thai Octogenarians
Record Dates: First submitted 2019-07-25; First posted 2019-08-07 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Stroke; Atrial Fibrillation
Keywords: anticoagulant drugs
MeSH Terms: conditions — Stroke; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non vitamin K oral anticoagulants (NOACs): Patients who were prescribed with apixaban, dabigatran, edoxaban, or rivaroxaban for stroke secondary prevention.
  Interventions: Drug: Non vitamin K oral anticoagulants
- Warfarin: Patients who were prescribed with warfarin for stroke secondary prevention.

INTERVENTIONS:
Drug: Non vitamin K oral anticoagulants — Non vitamin K oral anticoagulants are apixaban, dabigatran, rivaroxaban, and edoxaban
  Groups: Non vitamin K oral anticoagulants (NOACs)

SUMMARY:
A retrospective cohort study of Thai octogenarians with nonvalvular atrial fibrillation (NVAF) initiating apixaban, dabigatran, rivaroxaban or warfarin was conducted in medical school hospital in Thailand. Patients were recruited from January 1, 2013, to December 31, 2018. The efficacy outcome was early recurrence of stroke or transient ischemic attack (TIA) in 90 days after initiation of oral anticoagulants (OACs). The safety outcome were major bleeding and clinically relevant non-major bleeding complications in 180 days. Continuous variables were compared using independent t test and MannWhitney U test, and categorical variables were compared using chi-square test or Fisher's exact test. Furthermore, hazard ratios and P values were calculated by the use of multivariable Cox's regression analysis.

DETAILED DESCRIPTION:
This is a retrospective cohort study of Thai octogenarians with NVAF. Patients who were prescribed with apixaban, dabigatran, edoxaban, rivaroxaban or warfarin from January 1, 2013, to December 31, 2018 were recruited. The primary efficacy was recurrent ischemic stroke or TIA in 90 days after initiating OACs. The secondary efficacy were recurrent ischemic stroke or TIA in 180 days after initiating OACs. While any bleeding complications were defied as primary safety outcomes. Continuous variables were compared using independent t test and MannWhitney U test, and categorical variables were compared using chi-square test or Fisher's exact test.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 80 years old
* Patients who were diagnosed with I48, I63 or G45 from International Classification of Diseases 10th version (ICD-10). Patients who were diagnosed atrial fibrillation and flutter, cerebral infarction or transient cerebral ischemic attacks (TIA) and related syndromes)
* Patients were prescribed apixaban, dabigatran, edoxaban, rivaroxaban, or warfarin

Exclusion Criteria:

* Patients were prescribed oral anticoagulants for other indications

  1. Prophylaxis thromboembolic events in valvular atrial fibrillation
  2. Treatment of venous thromboembolism
  3. Prophylaxis thromboembolic events in hip or knee replacement
* Patients who had contraindication to oral anticoagulants

  1. Creatinine clearance calculated from Cockcroft-Gault equation 1.1 Creatinine clearance less than 30 mL/min (for patients who receiving Dabigatran) 1.2 Creatinine clearance less than 15 (mL/min (for patients who receiving Apixaban, Edoxaban, Rivaroxaban)
  2. Patients were diagnosed acute hepatitis, chronic active hepatitis

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Study Population: Patients aged over 80 years with non valvular atrial fibrillation who were prescribed oral anticoagulants (OACs) which were apixaban, dabigartran, edoxaban, rivaroxaban and warfarin for stroke secondary prevention.
Sampling Method: Non-Probability Sample
Enrollment: 327 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Rate recurrence of stroke or TIA in 90 days | 90 days after initiation of OACs
  Rate recurrence of stroke or TIA in 90 days after initiation of OACs

SECONDARY OUTCOMES:
Rate recurrence of stroke or TIA in 180 days | 180 days after initiation of OACs
  Rate recurrence of stroke or TIA in 180 days after initiation of OACs
Rate of major bleeding | 180 days after initiation of OACs
  Rate of major bleeding in 90 days and 180 days after initiation of OACs
Rate of clinically relevant non-major bleeding | 180 days after initiation of OACs
  Rate of clinically relevant non-major bleeding in 90 days and 180 days after initiation of OACs
Patients's baseline characteristics associated with recurrence of stroke or TIA as assessed by multivariate cohort analysis | 180 days after initiation of OACs
  Patients's baseline characteristics associated with recurrence of stroke or TIA in 180 days after initiation of OACs as assessed by multivariate cohort analysis
Patients's baseline characteristics associated with major bleeding and clinically relevant non-major bleeding as assessed by multivariate cohort analysis | 180 days after initiation of OACs
  Patients's baseline characteristics associated with major bleeding and clinically relevant non-major bleeding in 180 days as assessed by multivariate cohort analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Siriraj Hospital, Phramongkutklao Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
Primary outcome of this study